CLINICAL TRIAL: NCT01859819
Title: Reduced Burden of Oncologic Therapy in Advanced B-cell Lymphoma (REBOOT ABLY) in Children, Adolescents and Young Adults With CD20+ Mature B-Cell Lymphoma
Brief Title: Treatment for Advanced B-Cell Lymphoma
Acronym: REBOOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-157; L 10,753 (Other: New York Medical College)
Record Dates: First submitted 2013-04-16; First posted 2013-05-22 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diffuse Large Cell Lymphoma; Burkitt's Lymphoma; High Grade B-cell Lymphoma
Keywords: Pediatric; Lymphoma (NOT primary mediastinal B-cell lymphoma); B-Cell---Burkitt's like; Rituximab; Liposomal ARA-C
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group B (Experimental): De-novo Mature CD 20 + B-NHL excluding PMBL histology. Good Risk FAB Group B includes patients with St. Jude Stages I /II (unresected) and stage III/IV with diagnostic LDH <2 X ULN.
  REDUCTION: Cyclophosphamide, Vincristine, Prednisone, IT Methotrexate INDUCTION:Rituximab, Vincristine, Methotrexate, Leukovorin, Cyclophosphamide, Doxorubicin CONSOLIDATION: Rituximab, Methotrexate, Leukovorin, Cytarabine
  Interventions: Drug: Rituximab; Drug: IT Cytarabine
- Group C, CNS negative (Experimental): De-novo Mature CD 20 + B-ALL (> 25% Bone marrow blasts) without CNS involvement.
  REDUCTION: Cyclophosphamide, Vincristine, Prednisone, IT Methotrexate, IT Cytarabine INDUCTION: Rituximab, Vincristine, Methotrexate, Leukovorin, Cyclophosphamide, Doxorubicin, IT Methotrexate, IT Cytarabine CONSOLIDATION: Rituximab, Cytarabine, Etoposide MAINTENANCE: Vincristine, Prednisone, Methotrexate, Leukovorin, Cyclophosphamide, Doxorubicin, Etoposide, Cytarabine
  Interventions: Drug: Rituximab; Drug: IT Cytarabine
- Group C, CNS Positive (Experimental): De-novo Mature CD 20 + B-NHL with CNS involvement:
  1. Any L3 blasts in CSF
  2. Cranial nerve palsy (if not explained by extracranial tumor)
  3. Clinical spinal cord compression
  4. Isolated intracerebral mass
  5. Parameningeal extension: cranial and/or spinal REDUCTION: Cyclophosphamide, Vincristine, Prednisone, IT Methotrexate, IT Cytarabine INDUCTION: Rituximab, Methotrexate, Leukovorin, Cyclophosphamide, Doxorubicin, IT Methotrexate, IT Cytarabine, IT Liposomal ARA-C, Vincristine CONSOLIDATION: Rituximab, Cytarabine, Etoposide MAINTENANCE: Vincristine, Cyclophosphamide, Methotrexate, Leukovorin, Doxorubicin, IT Liposomal ARA-C,
  Interventions: Drug: Rituximab; Drug: IT Cytarabine

INTERVENTIONS:
Drug: Rituximab
  Other Names: RITUXAN®, IDEC-C2B8) NSC #687451, IND #10385
Drug: IT Cytarabine
  Other Names: DEPOCYT® (Cytarabine Liposome Injection)

SUMMARY:
To safely reduce the burden of therapy in children, adolescents and young adults with mature B-NHL by reducing the number of intrathecal (IT) injections by the introduction of IT Liposomal Cytarabine (L-ARA-C, [Depocyt®]) and reducing the dose of anthracycline (doxorubicin) in good risk patients with the addition of rituximab to the FAB chemotherapy backbone (Immunochemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed mature B-lineage (CD20 positive) Leukemia/Lymphoma
* 1. Diffuse Large Cell Lymphoma (NOT primary mediastinal B-cell lymphoma) -2. Burkitt's Lymphoma
* 3. High Grade B-cell Lymphoma---Burkitt's like.

B-Cell Anaplastic Large cell Ki 1 positive lymphomas, Primary Mediastinal B-Cell Lymphoma (PMBL), and B-Lymphoblastic lymphomas are ineligible.

No previous chemotherapy. Patients who have received emergency irradiation and/or steroid therapy will be eligible ONLY if started on protocol therapy not more than 72 hours from the start of radiotherapy or steroids. Bone marrow and cerebrospinal fluid MUST be obtained before steroids are given for patient to be eligible for the study.

Exclusion Criteria:

* Patients with newly diagnosed Group A (low risk) lymphoma. Patients with Group B (intermediate risk) if classified as Murphy Stage III/IV and diagnostic LDH > 2 XULN and patients with primary mediastinal B-cell lymphoma (PMBL).
* Patients who have received any steroids in the week prior to diagnosis except as stated in Section 4.1.4 of the protocol.
* No congenital or acquired immune deficiency. These patients are excluded due to the expected intense immunosuppression, increased risk of opportunistic infections, and higher expected septic death rate in this subgroup of patients with this proposed therapy.
* No prior solid organ transplantation.
* Patients with previous malignancies that have been treated with systemic chemotherapy with alkylator or anthracycline therapy. The latter group of patients are excluded due to an expected increase in late effects (eg. late cardiac toxicity, secondary malignancies, sterility, etc.).
* Patients with known G6PD deficiency are NOT ELIGIBLE for Rasburicase therapy. Patients with G6PD deficiency should be treated with alkalinization, IV hydration and po and/or IV allopurinol during the reduction phase (COP).

4.2.6 Patients with serious (sepsis, pneumonia, etc..) proven or suspected infections at diagnosis will be excluded.

4.2.7 Pregnancy or Breast-Feeding: No information is available regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 3 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
To determine if disease response rate will improve with this combination of therapy. | 1 year
  To determine if the addition of intrathecal ([IT] [Depocyt®]) and reduction of standard IT dosing and the reduction of anthracycline exposure (doxorubicin) (60%) within the ANHL01P1 FAB/LMB B4 + Rituximab chemoimmunotherapy backbone in children, adolescents and young adults with good risk CD20+ mature B-NHL (Stage I and II unresected and Stage III/IV with LDH < 2 UNL) will result in similar response rates compared to historical controls (Subgroup I).

SECONDARY OUTCOMES:
To determine if the combination of IT Depocyte®, Rituximab and FAB Chemotherapy is safe. | 1 year
  To determine the safety and efficacy of reduction of IT therapy and substitution with L-ARA-C (Depocyte®) within ANHL01P1 FAB/LMB Group C1 plus rituximab chemotherapy backbone in children, adolescents and young adults with advanced risk de-novo mature B-NHL (Group C BM±CNS) (Subgroup II) as measured by reported serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College; Stanton Goldman, MD, Study Director — Medical City Children's Hospital, Dallas
Locations (5):
- United States (5):
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Goldman S, Barth M, Shiramizu B, Shi Q, Hochberg J, Klejmont L, Harrison L, Basso J, Chu Y, Islam H, Gerard P, Agsalda-Garcia M, Shieh T, Oesterheld J, Heym K, Kirov I, Drachtman R, Harker-Murray P, Perkins S, Miles RR, Cairo M. A dose substitution of anthracycline intensity with dose-dense rituximab in children and adolescents with good-risk mature B-cell lymphoma. Leukemia. 2021 Oct;35(10):2994-2997. doi: 10.1038/s41375-021-01256-8. Epub 2021 May 3. No abstract available. PMID 33941850